CLINICAL TRIAL: NCT04503148
Title: The Influence of Type of Anesthesia on Recurrence of Renal Cell Carcinoma After Nephrectomy: a Prospective Randomized Controlled Study
Brief Title: Anesthesia and Cancer Study: Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ane-Can Nx
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Anesthesia; Propofol; Inhaled anesthetics; Renal cell carcinoma; Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Propofol; Anesthetics, Inhalation

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Experimental): Patients receiving the total intravenous anesthesia using propofol
  Interventions: Drug: Propofol
- inhalation group (Active Comparator): Patients receiving inhalation anesthesia using sevoflurane or desflurane
  Interventions: Drug: Inhaled General Anesthetics

INTERVENTIONS:
Drug: Propofol — Propofol 1-2 mg/kg bolus injection for induction of anesthesia propofol continuous infusion for maintenance of anesthesia
  Arms: TIVA group
Drug: Inhaled General Anesthetics — Sevoflurane or desflurane for induction and maintenance of anesthesia
  Arms: inhalation group

SUMMARY:
This study investigates the influence of type of anesthesia on recurrence and survival of renal cell carcinoma in patients undergoing nephrectomy. The participants will be allocated to either the group receiving the total intravenous anesthesia (TIVA) using propofol or the group receiving the inhaled anesthetics, such as sevoflurane or desflurane.

DETAILED DESCRIPTION:
The effect of anesthesia on cancer recurrence and survival is controversial. According to some retrospective studies and preclinical studies, TIVA is suggested to be more favorable than inhalation anesthesia regarding cancer recurrence and survival after surgery. However, to our knowledge, there is no study which investigates the influence of type of anesthesia on recurrence of renal cell carcinoma after nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for elective nephrectomy due to renal cell carcinoma

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Allergies to anesthetics
* Palliative surgery
* Refusal to participate in the study
* History of diagnosis or surgery for other cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
five year metastasis-free survival | five year after surgery
  five year metastasis-free survival

SECONDARY OUTCOMES:
one year survival | one year after surgery
  survival rate regardless of recurrence
three year survival | three year after surgery
  survival rate regardless of recurrence
one year metastasis-free survival | one years after surgery
  one year metastasis-free survival
three year metastasis-free survival | three years after surgery
  three year metastasis-free survival
five year survival | five year after surgery
  survival rate regardless of recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No